CLINICAL TRIAL: NCT03296371
Title: Genetics of Embryonal and Alveolar Rhabdomyosarcoma Study (GEARS)
Brief Title: Genetic Mutational Analysis of Saliva or Buccal Mucosa Samples From Patients With Embryonal or Alveolar Rhabdomyosarcoma
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AEPI15N1; NCI-2017-01665 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AEPI15N1 (Other: Childrens Oncology Group); AEPI15N1 (Other: CTEP)
Record Dates: First submitted 2017-09-19; First posted 2017-09-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Alveolar Rhabdomyosarcoma; Embryonal Rhabdomyosarcoma
MeSH Terms: conditions — Rhabdomyosarcoma, Alveolar; Rhabdomyosarcoma, Embryonal

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, buccal mucosa
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (biospecimen collection): Patients and their parents undergo collection of saliva or buccal mucosa samples for genetic mutational analysis. Germline DNA from saliva or buccal mucosa is evaluated via whole exome sequencing.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo saliva or buccal mucosa collection
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research trial studies genetic mutations in saliva or buccal mucosa samples from patients with embryonal or alveolar rhabdomyosarcoma. Identifying gene mutations may help doctors learn about the prognosis of patients with embryonal or alveolar rhabdomyosarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify novel recurrent de novo germline mutations among rhabdomyosarcoma (RMS) case-parent trios.

II. To identify the frequency of de novo germline mutations in cancer predisposition genes among RMS case-parent trios.

SECONDARY OBJECTIVES:

I. To conduct ?deep phenotyping? of children diagnosed with RMS utilizing questionnaire data and information from medical records.

OUTLINE:

Patients and their parents undergo collection of saliva or buccal mucosa samples for genetic mutational analysis. Germline deoxyribonucleic acid (DNA) from saliva or buccal mucosa is evaluated via whole exome sequencing.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be enrolled on ACCRN07 and/or APEC14B1 and registered with COG by a North American member institution
* The patient must have a diagnosis of embryonal rhabdomyosarcoma or alveolar rhabdomyosarcoma
* The patient must be diagnosed with rhabdomyosarcoma between January 1, 2012 and November 30, 2019
* Concomitant treatment on a therapeutic trial is not required
* The patient must have at least one biological parent alive and willing to participate
* All questionnaire respondents must understand English or Spanish
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with embryonal or alveolar rhabdomyosarcoma enrolled on ACCRN07 and/or APEC14B1 and registered with Children's Oncology Group (COG)
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2017-10-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Novel recurrent de novo germline mutation identification | Up to 3 years
  Will analyze de novo single-nucleotide variants (SNVs), copy-number variants (CNVs), and insertions/deletions (INDELs) obtained through next-generation exome sequencing of rhabdomyosarcoma (RMS) case-parent trios.
Frequency of de novo germline mutations in cancer predisposition genes | Up to 3 years
  Will conduct targeted sequencing using samples collected from the case and his/her parents in order to determine the prevalence of novel de novo mutations in cancer-syndrome genes associated with RMS.

SECONDARY OUTCOMES:
Deep phenotyping of children diagnosed with rhabdomyosarcoma utilizing questionnaires and medical record information | Up to 3 years
  Analyses will be descriptive in nature.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Lupo, Principal Investigator — Children's Oncology Group
Locations (1):
- Childrens Oncology Group, Philadelphia, Pennsylvania, United States